CLINICAL TRIAL: NCT06788925
Title: Clinical Evaluation of an Innovative Hypothermia Management Strategy in Trauma Patients: Effectiveness of the Therm'Up Heating Device
Brief Title: Clinical Evaluation of Effectiveness of the "Therm'Up" Heating Device
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: ThermoTrauma (Industry)
Collaborators: Digital Medical Hub (Other); Chambery Hospital, France (Unknown); Centre Hospitalier Annecy Genevois (Other); University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024-A02412-45
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Hypothermia Due to Cold Environment
Keywords: Hypothermia; Lifejacket; Active device
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm with ThermUp chest protector (Experimental): Patients benefi ting from the Therm'Up heated chest protector
  Interventions: Device: Patients support with active thermic jacket
- Control Arm with blanket (Active Comparator): Patients supported with survival coverage (conventional PEC).
  Interventions: Device: Patients support with survival coverage

INTERVENTIONS:
Device: Patients support with survival coverage — Following calls to emergency medical services, handled by the ground SMUR/SAMU or the air SMUR (HéliSMUR), the operator collects essential information on the nature of the incident and the apparent condition of the injured. A medical team is thus mobilized on site. It takes over from the rescue team (e.g. the SDIS fi refi ghters) who are generally the fi rst to arrive on the scene.
  Eligible patients will be randomly assigned consecutively to one of two groups: control (use of the survival blanket) and experimental (use of the Therm'Up breastplate).
  Any traumatized person at risk of hypothermia or in hypothermia in a pre-hospital environment, having given verbal consent to participate in the study and meeting the inclusion criteria
  Arms: Control Arm with blanket
Device: Patients support with active thermic jacket — The intervention Description is exactly the same, except that the patient will be given a ThermUp jacket
  Arms: Experimental Arm with ThermUp chest protector

SUMMARY:
Here's a concise summary in English without the numbers:

Hypothermia is defined as a core temperature below 35°C and occurs when the body loses more heat than it produces. It is classified by severity: mild (32-35°C), moderate (28-32°C), and severe (<28°C). Trauma patients are particularly vulnerable, as hypothermia can affect cardiac, pulmonary, neurological, and coagulation systems, contributing to the "lethal triad" of metabolic acidosis, coagulopathy, and hypothermia, which increases early mortality risk.

Shivering, a key sign of hypothermia, significantly raises oxygen consumption, making its prevention during prehospital care critical. Passive warming measures, such as insulating survival blankets, are commonly used to prevent heat loss in emergencies. These blankets help maintain body temperature, protecting victims from cold and wind. Hypothermia prevalence among trauma patients on hospital arrival is high, emphasizing the importance of prehospital measures to limit its impact. However, active warming systems are often impractical in prehospital settings, leaving passive methods as the primary strategy.

DETAILED DESCRIPTION:
Hypothermia is defi ned as a core temperature below 35°C. Accidental hypothermia occurs when the human body loses more heat than it produces, resulting in a drop in body temperature.

Core body temperature is the standard physiological parameter for diagnosing and classifying the severity of hypothermia. Mild accidental hypothermia is defi ned as a core body temperature between 32 and 35°C, moderate hypothermia as a core temperature between 28 and 32°C, and severe hypothermia as a core temperature <28°C.

Trauma patients are at high risk of accidental hypothermia (body temperature ≤ 35°C). Hypothermia has signifi cant consequences on human physiology, including the cardiac, pulmonary, neurological, and hemostatic systems.

Hypothermia is of particular concern in trauma patients because it is associated with increased morbidity and mortality. In addition, hypothermia can infl uence blood coagulation by reducing platelet aggregation and increasing fi brinolysis. Three closely related elements: metabolic acidosis, coagulopathy, and hypothermia constitute the "lethal triad" of trauma. The presence of one or more of these elements during the management of a severely traumatized patient increases the risk of early mortality.

The occurrence of shivering in a patient is also an indicator of hypothermia. Shivering can increase oxygen consumption of muscle cells by up to 400%. The goal of prehospital care is to prevent the onset of shivering, making the use of passive warming measures crucial.

In a systematic review, the prevalence of hypothermia in trauma victims on arrival at hospital was found to be high, at 14%.

An observational study conducted by the SMUR (Mobile Emergency and Resuscitation Services) team of eight French hospitals between January 1, 2004 and November 10, 2007, measured the body temperature of 448 patients upon arrival at the hospital. Hypothermia (body temperature ≤ 35°C) was present in 64 of these 448 patients (14%). Optimal patient care can help limit heat loss or hypothermia. It is important to note that the prolonged time required to recover patients after a road accident increases the risk of lasting hypothermia. This hypothermia, linked to the accident, is associated with an increased mortality rate in severely injured patients, which underlines the importance of prehospital efforts to prevent hypothermia.

Prevention of hypothermia in trauma patients in the prehospital care setting is of critical importance. Various devices have been designed to reduce heat loss and/or actively warm patients in a prehospital environment.

Warming strategies are not ideally suited to pre-hospital care due to the complexity of their implementation and their inadequacy to the conditions encountered. Active external systems generate heat transferred to the patient, while passive systems isolate the patient by preventing the dispersion of body heat.

In most cases, passive warming methods are used, such as the use of insulating survival blankets, which still allow the patient to be insulated from the cold. The insulating survival blanket is used in emergency situations to cover a victim and prevent hypothermia. It is an essential product in the event of illness or accident (trauma, fall, etc.), or in the event of a sudden change in temperature, to maintain the victim's body temperature, protect them from the cold and wind and prevent hypothermia. These so-called "isothermal" blankets allow the body temperature to be maintained at around 37°C.

Active external warming is only possible with chemical, electrical methods or warm air blankets, but these are diffi cult to access before arrival at the hospital due to their high cost, their signifi cant environmental impact (single use) and their unsuitability for outdoor use. However, only proactive and early administration of heat can effectively combat hypothermia and its consequences. The use of a heated blanket or better still, a warm air mattress, is much more effective and allows to gain 1 to 2 °C of core temperature per hour. In out-of-hospital and mountain rescue environments, measuring core temperature can guide transport and treatment decisions, although obtaining an accurate value can be difficult.

Developing alternatives to current devices would reduce health risks and allow targeted intervention to control core temperature, thereby preventing or reducing the harmful consequences of hypothermia. This type of innovation would also have the potential to reduce the risks and limitations associated with existing technical procedures. Hence the objective of this clinical investigation to assess the non-inferiority of a new Therm'Up device compared to the survival blanket to prevent hypothermia in trauma patients in prehospital care.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years; Confi dential Page 7on 11 Version No. 2.0 of 2024/12/10
* Patient at risk of hypothermia presenting with grade A, or B, or C trauma or patient with hypothermia;
* Patient exposed to cold;
* Patient with hemorrhage;
* Patient burned over 20% of body surface area;
* Patient requiring an intervention delay of more than 30 minutes (between the arrival of the medical team on site and arrival at the hospital)

Exclusion Criteria:

* Patient with known ongoing hyperthermia and/or infections or body injuries such as burns in the area where the breastplate is positioned;
* Patient presenting with cardiac arrest before the arrival of the team;
* Patient with bilateral aural bleeding preventing continuous monitoring of the eardrum;
* Patient covered with insulating bubble wrap;
* Pregnant or breastfeeding woman;
* Patient already participating in an interventional clinical trial;
* Patient not receiving social security benefi ts;
* Adult patient subject to a legal protection measure, guardianship or deprived of liberty by a judicial or administrative decision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-05 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Statistical distribution of the temperature evolution | From the intervention of the medical team on site until discharge from the hospital (1 month maximum)
  The statistical distribution of the temperature evolution will be tested to verify whether it follows a normal distribution. The Shapiro-Wilk test and graphical methods will be used to assess this normality.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Spadoni, Study Director — Thermotrauma SAS
Locations (1):
- Grenoble Alpes University Hospital, Échirolles, France

IPD SHARING:
Plan to Share IPD: No
According to European Regulation on Data Protection (GDPR, 2016/679, April 2016), we are not allowed to share patients data

REFERENCES:
- See also: Official website of the device (active jacket) — https://thermotrauma.com/